CLINICAL TRIAL: NCT06385626
Title: The Effects of Raspberry Leaf Tea on Blood Glucose Control in Healthy Adults
Brief Title: The Effects of Raspberry Leaf Tea on Blood Glucose Control
Acronym: RLT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Prof, University of Reading
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UREC: 23_15-Raspberry Leaf Tea
Record Dates: First submitted 2024-04-19; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Type II Diabetes
Keywords: glucose; polyphenols
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Volunteers will be asked to consume 50 g of carbohydrate powder (sucrose and glucose) with or without 10 g of raspberry leaf tea, which will be dissolved in 300 mL of warm water during four visits (every month).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- sucrose + raspberry leaf tea (Experimental): Volunteers will be asked to consume 50 g of sucrose with 10 g of raspberry leaf tea dissolved in 300 mL of warm water.
  Interventions: Dietary Supplement: Raspberry leaf tea
- glucose + raspberry leaf tea (Experimental): Volunteers will be asked to consume 50 g of glucose with10 g of raspberry leaf tea dissolved in 300 mL of warm water.
  Interventions: Dietary Supplement: Raspberry leaf tea
- sucrose (Active Comparator): Volunteers will be asked to consume 50 g of sucrose without 10 g of raspberry leaf tea
  Interventions: Dietary Supplement: Raspberry leaf tea
- glucose (Active Comparator): Volunteers will be asked to consume 50 g of glucose without 10 g of raspberry leaf tea
  Interventions: Dietary Supplement: Raspberry leaf tea

INTERVENTIONS:
Dietary Supplement: Raspberry leaf tea — 10 g of raspberry leaf tea

SUMMARY:
The aim of the present clinical trial is to assess how raspberry leaf polyphenols impact on postprandial glucose and insulin levels in healthy individuals consuming sucrose.

The questions the project will address:

* Do raspberry leaf polyphenols lower sucrose-induced increases in plasma glucose in humans?
* Do these polyphenols mediate these effects by inhibiting digestion of sucrose or the absorption of glucose.

  20 healthy adults will be recruited between the ages of 18-65 years who are non-smokers and not taking certain types of medication (e.g., drugs from a GP for high blood pressure, high blood fats, inflammatory conditions, and depression) or dietary supplements (e.g., cholesterol-lowering spreads, fish oil, probiotics, prebiotics, and natural laxatives), antibiotics in the last three months or if they used any drugs or supplements that could affect their blood glucose or lipid metabolism. No abnormal results for liver function tests, renal function tests, and lipid profile tests. If they have food allergies or consume more than 14 units of alcohol per week (i.e., to help they calculate a alcohol intake, one standard glass of wine (175 ml) or one pint of regular lager is equivalent to just over two units of alcohol), frequently travel for work or are participating in another intervention study, they will not be able to participate. Women who are pregnant or lactating or planning a pregnancy in the next six months will also not be able to take part, not use herbal medicines for at least the previous three months, not be on a weight loss program six months before screening, not involved in clinical trials six months before the screening, and not having severe cardiac, hepatic, or renal function impairment. Not Sufferers of chronic illnesses, not Individuals with food allergies, not people with coeliac disease.

They will be asked to attend a four-study visit after an eight-hour overnight fast. Volunteers will be asked to consume 50 g of carbohydrate powder (sucrose and glucose) with or without 10 g of raspberry leaf tea, which will be dissolved in 300 mL of warm water during four visits (every month). Blood samples will be taken at intervals for a period of two hours after the consumption of raspberry leaf or control. Blood glucose and insulin levels will be tested 15 minutes before, at 15,30,60,90, and 120 minutes after carbohydrate intake.

DETAILED DESCRIPTION:
The volunteer inclusion criteria are: (Fasting blood glucose in the range < 5.5 mmol/l (at day 0); A signed consent form; Age 18-65 years; Body mass index ≤ 34.9 kg/m2; Non-smoking; No pregnancy/lactation; No use of herbal medicines for at least the previous three months; Not on a weight loss program six months before screening; Not involved in clinical trial six months before screening; Not had severe cardiac, hepatic, or renal function impairment).

The volunteer exclusion criteria are: (Smoking, Pregnancy/lactation; Use of herbal medicines for at least the previous three months; Involved in a weight loss program six months before screening; Involved in clinical trial six months before the screening; Had severe cardiac, hepatic, or renal function impairment; Sufferers of chronic illnesses; Individuals with food allergies; People with prediabetes or diabetes; People with coeliac disease)

If all subjects are generally healthy, as demonstrated by their medical history and laboratory tests, including fasting blood sugar and insulin levels, as well as HOMA-IR, liver function tests (alanine transaminase, alkaline phosphatase, total bilirubin, and gamma-GT), renal function tests (uric acid and creatinine), and lipid profile tests (total cholesterol, Triglycerides). They will be asked to attend a four-study visit after an eight-hour overnight fast. Volunteers will be asked to consume 50 g of carbohydrate powder (sucrose and glucose) with or without 10 g of raspberry leaf tea, which will be dissolved in 300 mL of warm water during four visits (every month). Blood samples will be taken at intervals for a period of two hours after the consumption of raspberry leaf or control. Blood glucose and insulin levels will be tested 15 minutes before, at 15,30,60,90, and 120 minutes after carbohydrate intake.

ELIGIBILITY:
The volunteer inclusion criteria are:

* Fasting blood glucose in the range < 5.5 mmol/l (at day 0)
* A signed consent forms.
* Age 18-65 years
* Body mass index ≤ 34.9 kg/m2
* Non-smoking
* No pregnancy/lactation
* No use of herbal medicines for at least the previous three months
* Not on a weight loss program six months before screening
* Not involved in clinical trial six months before screening
* Not had severe cardiac, hepatic, or renal function impairment

The volunteer exclusion criteria are:

* Smoking
* Pregnancy/lactation
* Use of herbal medicines for at least the previous three months
* Involved in a weight loss program six months before screening.
* Involved in clinical trial six months before the screening.
* Had severe cardiac, hepatic, or renal function impairment.
* Sufferers of chronic illnesses
* Individuals with food allergies
* People with prediabetes or diabetes
* People with coeliac disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-12-23 (Estimated); Study Completion 2024-12-23 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose | Two hours
  Area under the plasma glucose curve 0-120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Spencer, PhD, Principal Investigator — University of Reading
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No